CLINICAL TRIAL: NCT06629558
Title: Efficacy and Safety of 0.5% w/v Nano- Silver Nitrate Versus Silver Nitrate Solution for Bronchoscopic Lung Volume Reduction in Management of Localized Emphysema: Prospective Interventional Randomized Controlled Clinical Trial
Brief Title: Bronchoscopic Lung Volume Reduction in Management of Localized Emphysema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer of chest medicine, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.24.09.2776
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Bronchoscopic Lung Volume Reduction
Keywords: bronchoscopic lung volume reduction; Nano-silver nitrate; Localized Emphysema; Silver nitrate
MeSH Terms: interventions — Silver Nitrate; Pneumonectomy; Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 0.5%w/v Nano- silver nitrate solution (Active Comparator): 0.5% weight by volume(w/v) Nano- silver nitrate solution for bronchoscopic lung volume reduction in management of localized emphysema
  Interventions: Drug: Nano-silver nitrate; Device: Bronchoscopic lung volume reduction
- 0.5%w/v silver nitrate solution (Active Comparator): 0.5%w/v silver nitrate solution for bronchoscopic lung volume reduction in management of localized emphysema
  Interventions: Drug: Silver Nitrate; Device: Bronchoscopic lung volume reduction

INTERVENTIONS:
Drug: Silver Nitrate — bronchoscopic lung volume reduction in management of localized emphysema
  Other Names: 0.5% w/v Silver nitrate solution
  Arms: 0.5%w/v silver nitrate solution
Drug: Nano-silver nitrate — bronchoscopic lung volume reduction in management of localized emphysema
  Other Names: 0.5% w/v Nano-silver nitrate solution
  Arms: 0.5%w/v Nano- silver nitrate solution
Device: Bronchoscopic lung volume reduction — bronchoscopic lung volume reduction in management of localized emphysema
  Other Names: Bronchoscopy

SUMMARY:
Emphysema is a progressive phenotype of chronic Obstructive Pulmonary Disease (COPD), poses a significant global health burden characterized by irreversible lung parenchymal destruction and airspace enlargement.

In recent years, bronchoscopic lung volume reduction (BLVR) has considerable interest as a minimally invasive approach to reducing hyperinflation and improving lung function in patients with emphysema.

BLVR techniques aim to achieve lung volume reduction by occluding or ablating emphysematous lung tissue through endobronchial delivery of various agents. Many techniques are available for BLVR as coil, endo-bronchial valve, and biological as thrombin, autologous blood and chemicals as silver nitrate solution.

DETAILED DESCRIPTION:
Emphysema is a progressive phenotype of chronic Obstructive Pulmonary Disease (COPD), poses a significant global health burden characterized by irreversible lung parenchymal destruction and airspace enlargement.

In recent years, bronchoscopic lung volume reduction (BLVR) has considerable interest as a minimally invasive approach to reducing hyperinflation and improving lung function in patients with emphysema.

BLVR techniques aim to achieve lung volume reduction by occluding or ablating emphysematous lung tissue through endobronchial delivery of various agents. Many techniques are available for BLVR as coil, endo-bronchial valve, and biological as thrombin, autologous blood and chemicals as silver nitrate solution.

Chemical lung volume reduction is an endo-bronchial approach, which uses chemical agents aiming to reduce lung volume by blocking off the most emphysematous areas with a rapidly polymerizing sealant. Endobronchial Valves (EBVs) show an overall success rate of 70-80% in reducing lung volume and improving lung function. Lung volume reduction coils (LVRC-Coils) have a success rate of 50-60%.

Bronchoscopic lung volume reduction with silver nitrate as a chemical agent was used in previous studies using a concentration of 0.5% and showed significant improvement in forced expiratory volume in first second (FEV1), diffusion capacity of lung to carbon monoxide (DLCo), modified Medical Research Council (mMRC) score when compared to base line values and reduction of the High Resolution Computed Tomography (HRCT) volumetry of the emphysematous regions.

Silver nanoparticles (AgNPs) are the most widely used nanomaterial today. These have found a wide range of applications in various areas such as textiles, agriculture, renewable energy, food, catalysis, bioremediation, and biomedicine

ELIGIBILITY:
Inclusion Criteria:

* COPD of grade III and IV according to GOLD 2024 staging of COPD with localized (heterogeneous) emphysema as determined by high resolution computerized tomography (HRCT) of the chest with area of destruction >-950 Hounsfield units (HU) and respiratory symptoms despite optimal medical therapy with the following criteria: Patient less than 75 years of age not candidate for or had refused lung volume reduction surgery but fit for fibro-optic bronchoscope (FOB). Lung volumes criteria: FEV1 less than 60% of predicted value, Residual volume (RV) more than 100% of predicted value, Total lung capacity (TLC) more than 100% of predicted value, 6 MWT of less than 450 meters.

Exclusion Criteria:

* Significant co-morbidities that limits exercise capacity or prognosis as cardiovascular diseases (heart failure, arrhythmia, ischemic heart disease) and lung cancer.
* Patients unfit or refused FOB.
* Homogenous emphysema.
* More than 75 years of age.
* Associated lung fibrosis.
* FEV1 > 60%.
* Current smoker.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Residual volume/ Total lung capacity (RV/TLC) ratio and volumetry | 6 months
  RV/TLC ratio measured at 6 months following treatment. Treatment success is defined as a statistically significant reduction in RV/TLC and from baseline.
change in Forced expiratory volume at first second (FEV1) and Forced vital capacity (FVC) | 6 months
  change from baseline to 6 months in FEV1 and FVC,
Voluometry | 6 months
  Voluometry measured at 6 months following treatment. Treatment success is defined as a statistically significant reduction in voluometry and from baseline.
diffusing capacity of the lung for carbon monoxide (DLCO) | 6 months
  change from baseline to 6 months in diffusing capacity of the lung for carbon monoxide (DLCO)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Mansoura University
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt